CLINICAL TRIAL: NCT03438123
Title: A Prospective Data Collection Study for the Evaluation of Performance and Safety of the Spectrum Dynamics Multi-purpose CZT SPECT Camera
Brief Title: Data Collection Study for the Spectrum Dynamics Multi-purpose CZT SPECT Camera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrum Dynamics (Industry)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SD-MPC-01
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Dementia; Parkinson Disease; Pulmonary Hypertension; Heart Diseases; Paget Disease; Bone Diseases; Bone Fracture; Renal Disease; Pulmonary Embolism; Bone Lesion
MeSH Terms: conditions — Dementia; Parkinson Disease; Hypertension, Pulmonary; Heart Diseases; Bone Diseases; Fractures, Bone; Kidney Diseases; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: All subjects undergo baseline clinically referred routine nuclear scintigraphy imaging and sequential imaging on the CZT SPECT investigational device following a single dose of radiopharmaceutical. Some subjects will additionally undergo CT on the CZT SPECT-CT investigational device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CZT SPECT (Experimental): CZT SPECT imaging with/without the addition of CT on the Spectrum Dynamics camera
  Interventions: Device: CZT SPECT imaging

INTERVENTIONS:
Device: CZT SPECT imaging — Acquisition of SPECT (single photon emission computed tomography) imaging utilising a camera system with solid-state cadmium zinc telluride (CZT) detectors to visualise injected, or otherwise introduced, radioactivity in the human body.

SUMMARY:
This study evaluates SPECT image data acquired from Spectrum Dynamics' multi-purpose CZT SPECT-CT camera. All subjects will undergo routine clinical Anger SPECT imaging and an additional SPECT acquisition on the CZT SPECT camera. Additionally some subjects will undergo CT on the CZT SPECT-CT camera. The quality of images from each device will be compared.

DETAILED DESCRIPTION:
The Spectrum Dynamics Multi-purpose CZT SPECT camera is a whole body SPECT (single photon emission computed tomography) scanner which utilises solid-state cadmium zinc telluride (CZT) detectors to visualise injected, or otherwise introduced, radioactivity in the human body. The CZT SPECT camera detects the location and distribution of gamma-emitting radionuclides in the body and produces 3 dimensional cross-sectional images through computed reconstruction of the data for the purpose of determining various metabolic and physiologic functions in the human body. In comparison to conventional sodium iodide (NaI) gamma camera (or Anger camera) technology, solid state CZT technology offers improved energy, spatial and temporal resolution, and higher count rates. Improvements in energy resolution and sensitivity thus enable the potential capability for enhanced quantification, simultaneous dual isotope imaging and dynamic imaging acquisition. The camera system also incorporates a multi-slice CT gantry and acquired SPECT and CT images can be combined to improve image reconstruction by allowing fusion of CT and SPECT image data for anatomic localisation referencing and CT attenuation correction of the SPECT image data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is clinically referred for scintigraphy using a radiopharmaceutical in the energy range of 40 - 220 keV emission
2. Patient is aged ≥18 years
3. Patient condition is stable
4. Patient is willing and able to undergo image acquisition on the MPC CZT SPECT camera with integrated CT in addition to standard clinical scintigraphy procedure
5. Patient must be willing and able to provide written informed consent
6. Patient must be affiliated to a social security scheme

Exclusion Criteria:

1. Patient with unstable medical condition
2. Patient is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
3. Patient is contra-indicated to undergo the scintigraphy imaging procedure for which they have been clinically referred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
CZT SPECT Image Acquisition | 1 day
  Technical adequacy of acquired CZT SPECT images for demonstrating the location and distribution of gamma ray radionuclides within the body
CZT SPECT-CT Image Acquisition | 1 day
  Technical adequacy of acquired CZT SPECT-CT images for demonstrating the location and distribution of gamma ray radionuclides within the body

SECONDARY OUTCOMES:
CZT SPECT Image Quality | 1 day
  Quality of acquired SPECT images from the CZT SPECT camera
Comparative Quality of CZT and Anger SPECT Images | 1 day
  Quality of acquired CZT SPECT images in comparison to the quality of images obtained from a conventional Anger gamma camera
Safety of the CZT SPECT Camera | Through study completion; anticipated to be 24 months
  Incidence of device related Adverse Events occurring during clinical use of the Spectrum Dynamics Multi-purpose CZT SPECT camera
Safety of the CZT SPECT Camera During Imaging Procedures | 1 day
  Incidence of peri-procedural Adverse Events
CZT SPECT-CT Image Quality | 1 day
  Quality of acquired SPECT-CT images from the CZT SPECT-CT camera
Comparative Quality of CZT SPECT-CT and Anger SPECT Images | 1 day
  Quality of acquired CZT SPECT-CT images in comparison to the quality of images obtained from a conventional Anger gamma camera
Safety of the CZT SPECT-CT Camera | Through study completion; anticipated to be 24 months
  Incidence of device related Adverse Events occurring during clinical use of the Spectrum Dynamics Multi-purpose CZT SPECT-CT camera
Safety of the CZT SPECT-CT Camera During Imaging Procedures | 1 day
  Incidence of peri-procedural Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Denis Agostini, MD.PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No